CLINICAL TRIAL: NCT03355079
Title: Efficacy of Long-term Parenteral Nutrition With SmofKabiven® E Concomitant to Chemo- and/or Immunotherapy: A Prospective, Randomised, Controlled, Open, Multicentre, Two-stage, Adaptive Clinical Trial in Metastatic Non-small Cell Lung Cancer
Brief Title: Efficacy Study of Long-term Parenteral Nutrition With SmofKabiven® E in Lung Cancer Patients Under Anticancer Therapy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low Patient Recruitment
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SMKV-013-CP4
Record Dates: First submitted 2017-11-16; First posted 2017-11-28 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Cancer-related Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SmofKabiven® E + standard oral nutrition (Experimental): SmofKabiven® E, with or without addition of Suppliven®, Vitalipid® Adult and/or Soluvit® will be administered at 5-7 days per week for up to 9 +/-1 weeks in addition to standard of care oral nutrition as per routine dietary counseling, to reach the patient's target energy intake.
  Interventions: Drug: SmofKabiven® E
- Standard oral nutrition (No Intervention): The patients will consume standard of care oral nutrition as per routine dietary counseling, to reach their target energy intake. Standard of care tube feeding or parenteral nutrition is allowed to start earliest 3 weeks after baseline visit, if required.

INTERVENTIONS:
Drug: SmofKabiven® E — In the intervention arm, SmofKabiven® E, with or without addition of Suppliven®, Vitalipid® Adult and/or Soluvit®, will be administered in addition to standard of care oral nutrition as per dietary counseling, whereas in the control arm, oral nutrition as per dietary counseling is the primary nutritional support.
  Arms: SmofKabiven® E + standard oral nutrition

SUMMARY:
The purpose of this study is to determine the efficacy of long-term addition of SmofKabiven® E to normal oral nutrition after routine dietary counseling as compared to standard of care nutrition in which oral nutrition is the primary nutritional support. It takes place in lung cancer patients under chemo- and/or immunotherapy. Efficacy will be determined primarily by calculating the change of patient's body weight from before start of study treatment to end of treatment, and comparing this change between both treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic non-small cell lung cancer patient
* Adult ≥ 18 years
* Starting any 1st, 2nd or 3rd line chemotherapy and/or immunotherapy administered via a central venous catheter (including implanted ports), or receiving the 2nd cycle of aforementioned anticancer treatment
* An energy gap of ≥ 40 % and/or 1000 kcal between the target energy intake (30 ± 5 kcal/kg/day) and the actual energy intake at screening, irrespective of weight loss
* Functional digestive tract allowing oral intake
* If female of childbearing potential, willing to use a sufficiently safe contraception method throughout participation in the study
* Signed informed consent from patient or legal representative

Exclusion Criteria:

* Parenteral nutrition (PN) administered during the preceding month (the sole administration of intravenous glucose is allowed), or standard of care PN planned to start within 3 weeks after baseline visit
* More than 1600 kcal/day required as PN
* Tube feeding at screening, or planned to start within 3 weeks after baseline visit
* Body mass index (BMI) > 30 kg/m2
* Performance status > 3 Eastern Cooperative Oncology Group (ECOG) score
* Life expectancy < 3 months
* Active bloodstream infection demonstrated by positive blood culture at Screening
* Hypersensitivity to fish-, egg, soya- or peanut protein or to any of the active substances or excipients in SmofKabiven E
* Severe blood coagulation disorders
* Congenital errors of amino acid metabolism
* Pathologically elevated serum levels of any of the included electrolytes
* General contraindications to infusion therapy: acute pulmonary oedema, hyperhydration, decompensated cardiac insufficiency
* Hemophagocytotic Syndrome
* Severe hyperlipidemia (serum triglycerides > 353 mg/dL)
* Severe liver insufficiency: liver enzymes (aspartate aminotransferase [AST], alanine aminotransferase [ALT], gamma glutamyl transferase [GGT]) or conjugated bilirubin exceeding 3 x upper limit of normal range, or International Normalised Ratio (INR) > 2
* Severe renal dysfunction (estimated glomerular filtration rate [eGFR] < 30 ml/min/1.73m2) and patients on renal replacement therapy
* Uncontrolled hyperglycaemia
* Unstable conditions (e.g., embolism, metabolic acidosis, hypotonic dehydration)
* Pregnancy or lactation
* Contraindications to any of the study assessment methods including computer tomography and indirect calorimetry
* Participation in a clinical study with an investigational drug or investigational medical device within one month prior to start of study or during study
* Prior inclusion in the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Change in total body weight (kg) | Every 2-3 weeks, for up to 9 +/-1 weeks

SECONDARY OUTCOMES:
Serum albumin | Every 2-3 weeks from baseline to final visit at 9 +/1 weeks after baseline
Serum transthyretin | Every 2-3 weeks from baseline to final visit at 9 +/1 weeks after baseline
Nutritional Risk Index | Every 2-3 weeks from baseline to final visit at 9 +/1 weeks after baseline
Unplanned PN or tube feeding according to standard of care in control group | Every 2-3 weeks from baseline to final visit at 9 +/1 weeks after baseline
Early termination of PN due to improvement in test group | Every 2-3 weeks from baseline to final visit at 9 +/1 weeks after baseline
Lean body mass determined from computer tomography (CT) scan at 3rd lumbar vertebra | Baseline to final visit at 9 +/1 weeks after baseline
Optional: lean tissue mass, phase angle and hydration status including intra- and extracellular body water with bioelectrical impedance analysis (BIA), if BIA device is available. | Baseline to final visit at 9 +/1 weeks after baseline
Karnofsky performance status | Every 2-3 weeks from baseline to final visit at 9 +/1 weeks after baseline
ECOG performance status | Time Frame: Every 2-3 weeks from baseline to final visit at 9 +/1 weeks after baseline
Handgrip strength in kg, using hand dynamometer | Every 2-3 weeks from baseline to final visit at 9 +/1 weeks after baseline
Actual and target number of completed chemotherapy and/or immunotherapy cycles | Every 2-3 weeks from baseline to 3 months after baseline
Actual dose and target chemotherapy and/or immunotherapy dose administered | Every 2-3 weeks from baseline to 3 months after baseline
Chemotherapy and/or immunotherapy toxicities according to NCI-CTC v4.0 including dose-limiting toxicities | Every 2-3 weeks from baseline to final visit at 9 +/1 weeks after baseline
Fatigue using the brief fatigue inventory (BFI questionnaire) | Every 2-3 weeks from baseline to final visit at 9 +/1 weeks after baseline
Overall survival | Until 6 months post baseline
Progression-free survival | At 3 and 6 months post baseline
Partial response rate (as per RECIST v 1.1) | At 9 +/-1 weeks, 3 months and 6 months after baseline
Complete response rate (as per RECIST v 1.1) | At 9 +/-1 weeks, 3 months and 6 months after baseline
Unplanned hospitalization | From baseline until 6 months after baseline
Quality of life (Functional Assessment of Cancer Therapy- General [FACT-G] score) | From baseline until final visit at 9 +/-1 weeks after baseline
Number of patients terminating anti-cancer and nutrition therapy as part of end-of-life care | From baseline until final visit at 9 +/-1 weeks after baseline
Resting energy expenditure | From baseline until final visit at 9 +/-1 weeks after baseline
  measured by indirect calorimetry
Ocurrence of unplanned admission to nursing home | From baseline until final visit at 9 +/-1 weeks after baseline

OTHER OUTCOMES:
Aspartate Aminotransferase | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Alanine Aminotransferase | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Alkaline phosphatase | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Gamma-Glutamyl Transferase | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Direct bilirubin | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Total bilirubin | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Internal Normalized Ratio | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Serum creatinine | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Serum urea | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Serum sodium | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Serum potassium | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Serum total calcium | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Serum magnesium | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Serum chloride | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Serum phosphate | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Serum bicarbonate | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Serum glucose | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Serum triglycerides | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Red blood cell count | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Total white blood cell count | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Differential blood count | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Haemoglobin | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Haematocrit | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Platelet count | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
C-reactive protein | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Blood pressure | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Heart rate | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Body temperature | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline
Infection rate including catheter-related blood stream infections demonstrated by positive blood culture | From baseline every 2-3 weeks until final visit at 9 +/-1 weeks after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Durand, MD, Principal Investigator — Hôpital Cochin, Paris
Locations (1):
- Hôpital Cochin, Paris, France